CLINICAL TRIAL: NCT04811664
Title: A Randomized Controlled Study to Assess SARS CoV-2 Infection, Viral Shedding, and Subsequent Potential Transmission in Individuals Immunized With Moderna COVID-19 Vaccine
Brief Title: A Study of SARS CoV-2 Infection and Potential Transmission in Individuals Immunized With Moderna COVID-19 Vaccine
Acronym: CoVPN 3006
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: CoVPN 3006
Record Dates: First submitted 2021-03-19; First posted 2021-03-23 (Actual); Results first posted 2023-07-27 (Actual); Last update posted 2023-08-02 (Actual); Status verified 2023-07

CONDITIONS: SARS-CoV-2 Infection
Keywords: SARS-CoV-2
MeSH Terms: conditions — COVID-19 | interventions — 2019-nCoV Vaccine mRNA-1273

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Immediate Vaccination (Experimental): Participants will receive Moderna COVID-19 Vaccine in 100 mcg dose given as 0.5 ml Intramuscular into the deltoid muscle on Day 1 and Day 29.
  Interventions: Biological: Moderna COVID-19 Vaccine
- Standard of care (Experimental): Participants will receive Moderna COVID-19 Vaccine in 100 mcg dose given as 0.5 ml Intramuscular into the deltoid muscle on Day 113 and Day 141.
  Interventions: Biological: Moderna COVID-19 Vaccine
- Vaccine Declined (No Intervention): Participants who prefer not to be vaccinated, If requested, participant will be offered vaccine if they have not received vaccine outside of the study

INTERVENTIONS:
Biological: Moderna COVID-19 Vaccine — A lipid nanoparticle (LNP) dispersion of a messenger ribonucleic acid (mRNA) encoding the prefusion stabilized S protein of SARS-CoV-2 formulated in LNPs composed of 4 lipids (1 proprietary and 3 commercially available). It is a suspension for intramuscular injection administered as a series of two doses (0.5 mL each) 1 month apart.
  Other Names: mRNA-1273
  Arms: Immediate Vaccination; Standard of care

SUMMARY:
The purpose of this study is to assess SARS CoV-2 infection, viral shedding, and subsequent potential transmission in individuals immunized with the Moderna COVID-19 vaccine.

DETAILED DESCRIPTION:
This study will evaluate the efficacy of the Moderna COVID-19 vaccine against SARS-CoV-2 infection, as well as its effect on peak nasal viral load as a measure of infection and a proxy of infectiousness, in adults aged 18-29.

In the Main study, up to 12,000 participants will be randomized 1:1 to Immediate Vaccination Group 1 (at Months 0 and 1) or Standard of Care Group 2, with vaccination given at Months 4 and 5 if not received off-study previously. Up to an additional 6,000 participants will be enrolled into the Vaccine Declined Group 3 and will also be offered vaccine at Months 4 and 5.

Additional study visits for Group 1 will occur at Months 2 and 4; for Groups 2 and 3, at Months 0 and 2. Study visits may include medical history, vaccine injections, blood collection, nasal swab, SARS-CoV-2 screening, COVID-19 symptom check, and questionnaires.

In addition to the main study participants, the study will also evaluate infectiousness following close contacts with main study participants. Study procedures for close contacts include questionnaires and blood samples; for those who become SARS-CoV-2 infected, study procedures will also include nasal swabs.

ELIGIBILITY:
Inclusion criteria for Main cohort, Vaccine Declined Group General and Demographic Criteria

* Age of 18 through 29 years.
* Ability and willingness to provide informed consent.
* Prefers not to receive COVID-19 vaccine.
* Willingness to be followed for the planned duration of the study.
* Assessment of understanding: volunteer demonstrates understanding of this study; completes a questionnaire with demonstration of understanding of all questionnaire items answered incorrectly.
* Access to device and internet for completion of study procedures.

Exclusion criteria for Main cohort, Vaccine Declined Group

* Prior administration of a coronavirus (SARS-CoV-2, SARS-CoV, MERS-CoV) vaccine or current/planned simultaneous participation in another interventional study to prevent or treat COVID-19 (participation in studies of other investigational research agents allowed).
* Any medical, psychiatric, occupational, or other condition that, in the judgment of the investigator, would interfere with, or serve as a contraindication to, protocol adherence, or a volunteer's ability to give informed consent.

Inclusion criteria for Prospective Close Contact (PCC) cohort

* Age of 18 years or older, at the time of signing the informed consent.
* Willing and able to provide informed consent.
* Expected to be in frequent close physical proximity with Main Cohort participant during the study.
* Willing to share results of SARS-CoV-2 testing.
* Access to device and internet for completion of study procedures

Inclusion criteria for Case-ascertained Close Contact (CACC) cohort

* Age of 18 years or older, at the time of signing the informed consent.
* Willing and able to provide informed consent.
* Access to device and internet for completion of study procedures.
* Willing to share results of SARS-CoV-2 testing.
* Had close contact with Main Cohort participant with known PCR-confirmed SARS-CoV-2 infection (eg, index case). Close contacts will have had exposure to the index participant, generally within 72 hours of an index diagnosis, and may include individuals that meet any of the following guidelines:

Prolonged close physical proximity with Main Cohort participant within a residence/vehicle/enclosed space without maintaining social distance,

Medical staff, first responders, or other care persons who cared for the index case without appropriate personal protective equipment.

Further information on the definition of close contact can be found in the CoVPN 3006 Study Specific Procedures (SSP).

Ages: 18 Years to 29 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1923 (Actual)
Dates: Start 2021-03-24 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2021-12-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn Stephenson, Study Chair — Harvard University School of Medicine; Audrey Pettifor, Study Chair — Gillings School of Global Public Health, University of North Carolina; Jasmine Marcelin, Study Chair — University of Nebraska
Locations (51):
- United States (51):
  - Alabama CRS, Birmingham, Alabama
  - Headlands Research Scottsdale, Scottsdale, Arizona
  - AMR Phoenix, Tempe, Arizona
  - University of Arizona, Tucson, Arizona
  - Charles Drew University, Los Angeles, California
  - UC Davis, Sacramento, California
  - University of California, San Diego, San Diego, California
  - University of Colorado- Boulder, Boulder, Colorado
  - JEM Headlands LLC, Atlantis, Florida
  - University of Florida, Gainesville, Florida
  - UF CARES, Jacksonville, Florida
  - Orlando Immunology Center CRS, Orlando, Florida
  - Headlands Research Sarasota, Sarasota, Florida
  - University of South Florida, Tampa, Florida
  - Morehouse University, Atlanta, Georgia
  - The Hope Clinic of the Emory Vaccine Center CRS, Decatur, Georgia
  - Champaign-Urbana Public Health District, Champaign, Illinois
  - Rush University CRS, Chicago, Illinois
  - Northwestern University, Evanston, Illinois
  - Indiana University, Bloomington, Indiana
  - Univ, of Kansas School of Medicine CRS, Wichita, Kansas
  - University of Kentucky, Lexington, Kentucky
  - Centex Studies, Inc. - Lake Charles, Lake Charles, Louisiana
  - University of Maryland College Park, College Park, Maryland
  - Fenway Health (FH) CRS, Boston, Massachusetts
  - Wayne State - Harper Hospital, Detroit, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - Columbia - Missouri VTEU, Columbia, Missouri
  - Washington University Therapeutics CRS, St Louis, Missouri
  - University of Nebraska, Omaha, Nebraska
  - AMR Las Vegas, Las Vegas, Nevada
  - University of New Mexico, Albuquerque, New Mexico
  - NYU Long Island Vaccine Center, Mineola, New York
  - NYU Bellevue Vaccine Center, New York, New York
  - Harlem Prevention Center CRS, New York, New York
  - New York Blood Center CRS, New York, New York
  - Stony Brook University, Stony Brook, New York
  - Bronx Prevention Research Center CRS, The Bronx, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - Wake Forest University, Winston-Salem, North Carolina
  - The Miriam Hopsital CRS, Providence, Rhode Island
  - Clemson University, Clemson, South Carolina
  - Vanderbilt Vaccine CRS, Nashville, Tennessee
  - Texas Tech, Amarillo, Texas
  - Centex Studies, Inc. - Brownsville, Brownsville, Texas
  - Texas A&M University, College Station, Texas
  - Centex Studies, Inc. - Houston, Houston, Texas
  - Centex Studies, Inc. - Westfield, Houston, Texas
  - Texas A&M - Kingsville, Kingsville, Texas
  - University of Virginia, Charlottesville, Virginia
  - University of Washington, Seattle, Washington

REFERENCES:
- [Derived] Vielot NA, Kelly NK, Ludema C, Rosenberg M, Brown ER, Janes HE, Kublin JG, Stephenson KE, Marcelin JR, Pettifor A. Patterns and predictors of COVID-19 vaccination among young adults at 44 US sites: Secondary analysis of a randomized, controlled, open-label trial, March - December 2021. Vaccine. 2024 Oct 3;42(23):126237. doi: 10.1016/j.vaccine.2024.126237. Epub 2024 Aug 24. PMID 39182315
- [Derived] Stephenson KE, Marcelin JR, Pettifor AE, Janes H, Brown E, Neradilek M, Yen C, Andriesen J, Grunenberg N, Espy N, Trahey M, Fischer RSB, DeSouza CA, Shisler JL, Connick E, Houpt ER, Chu HY, McCulloh RJ, Becker-Dreps S, Vielot NA, Kalbaugh CA, Cherabuddi K, Krueger KM, Rosenberg M, Greenberg RN, Joaquin A, Immergluck LC, Corey L, Kublin JG. Efficacy of Messenger RNA-1273 Against Severe Acute Respiratory Syndrome Coronavirus 2 Acquisition in Young Adults From March to December 2021. Open Forum Infect Dis. 2023 Nov 2;10(11):ofad511. doi: 10.1093/ofid/ofad511. eCollection 2023 Nov. PMID 38023544

RESULTS

PARTICIPANT FLOW:
Groups:
- Immediate Vaccination: Immediate Vaccination Group: Participants will receive Moderna COVID-19 Vaccine in 100 mcg dose given as 0.5 ml Intramuscular into the deltoid muscle on Day 1 and Day 29.
- Standard of Care: Standard of Care Group: Participants will receive Moderna COVID-19 Vaccine in 100 mcg dose given as 0.5 ml Intramuscular into the deltoid muscle on Day 113 and Day 141.
- Vaccine Declined: Vaccine Declined: Participants who prefer not to be vaccinated, If requested, participant will be offered vaccine if they have not received vaccine outside of the study
Period: Overall Study
Arm/Group | Immediate Vaccination | Standard of Care | Vaccine Declined
Started | 725 | 728 | 470
Full Analysis Set (FAS) | 725 | 728 | 470
Full Analysis Set With Study PCR (FAS-P) | 701 | 646 | 454
FAS-P With Outside Vaccination Censored Incidence Rate Follow-up | 563 | 622 | 452
Baseline Negative | 600 | 549 | 311
Baseline Negative With Outside Vaccination Censored Incidence Rate Follow-up | 489 | 531 | 311
FAS-P Viral Load | 22 | 23 | 44
Completed | 571 | 450 | 255
Not Completed | 154 | 278 | 215
Not completed — Lost to Follow-up | 78 | 125 | 46
Not completed — Withdrawal by Subject | 39 | 76 | 12
Not completed — Participant Unable to Adhere to Visit Schedule | 6 | 13 | 17
Not completed — Participant is unwilling or unable to comply with required study | 24 | 47 | 16
Not completed — Protocol Violation | 0 | 5 | 11
Not completed — Study Terminated by Sponsor | 4 | 3 | 34
Not completed — Early Study Closure | 3 | 7 | 79
Not completed — Other (Unable to receive payment visa status) | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Population: Baseline Negative
Groups:
- Total: Total of all reporting groups
Arm/Group | Immediate Vaccination | Standard of Care | Vaccine Declined | Total
Number analyzed (Participants) | 600 | 549 | 311 | 1460
Age, Continuous [Median (Full Range); unit: years] | 21 [18 to 29] | 21 [18 to 29] | 22 [18 to 29] | 21 [18 to 29]
Age, Customized [Count of Participants; unit: Participants]
  18 - 22 years | 449 | 402 | 157 | 1008
  23 - 26 years | 122 | 128 | 84 | 334
  27 - 29 years | 29 | 19 | 70 | 118
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Man | 254 | 248 | 126 | 628
  Woman | 321 | 282 | 175 | 778
  Transgender Man | 3 | 1 | 1 | 5
  Transgender Woman | 0 | 1 | 0 | 1
  Gender Nonconforming/Gender Variant | 3 | 7 | 3 | 13
  Genderqueer | 3 | 1 | 0 | 4
  Other | 1 | 2 | 1 | 4
  Multiple | 10 | 7 | 1 | 18
  Unknown | 5 | 0 | 4 | 9
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 341 | 294 | 184 | 819
  Male | 259 | 255 | 127 | 641
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: Because some participants did not report the characteristic sum of Ns across categories is less than the Overall Number of Baseline Participants.
  Participants
    number analyzed (Participants) | 596 | 547 | 308 | 1451
    Hispanic or Latino | 106 | 99 | 71 | 276
    Not Hispanic or Latino | 490 | 448 | 237 | 1175
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 3 | 1 | 6
  Asian | 97 | 93 | 11 | 201
  Native Hawaiian or Other Pacific Islander | 2 | 1 | 1 | 4
  Black or African American | 47 | 49 | 47 | 143
  White | 358 | 334 | 203 | 895
  More than one race | 52 | 43 | 26 | 121
  Other | 19 | 13 | 8 | 40
  Prefer not to answer | 23 | 13 | 14 | 50
Region of Enrollment [Count of Participants; unit: Participants]
  USA | 600 | 549 | 311 | 1460
Residence [Count of Participants; unit: Participants] — Population: Because some participants did not report the characteristic sum of Ns across categories is less than the Overall Number of Baseline Participants.
  Participants
    number analyzed (Participants) | 600 | 549 | 310 | 1459
    Dormitory or campus housing | 87 | 78 | 21 | 186
    Fraternity or sorority house | 9 | 10 | 0 | 19
    Apartment building or condo | 285 | 258 | 146 | 689
    Stand-alone house (non-fraternity or sorority) | 190 | 178 | 128 | 496
    Shelter | 0 | 1 | 2 | 3
    RV / Trailer | 4 | 3 | 3 | 10
    Staying with friends / Couch surfing | 4 | 3 | 2 | 9
    No residence | 0 | 0 | 2 | 2
    Other | 21 | 18 | 6 | 45
Number of roommates (sleep in same room) [Count of Participants; unit: Participants] — Population: Because some participants did not report the characteristic sum of Ns across categories is less than the Overall Number of Baseline Participants.
  Participants
    number analyzed (Participants) | 599 | 548 | 308 | 1455
    0 | 392 | 362 | 150 | 904
    1 | 170 | 157 | 124 | 451
    >1 | 37 | 29 | 34 | 100
Number of people in shared communal space [Count of Participants; unit: Participants] — Population: Because some participants did not report the characteristic sum of Ns across categories is less than the Overall Number of Baseline Participants.
  Participants
    number analyzed (Participants) | 599 | 548 | 308 | 1455
    0 | 66 | 63 | 37 | 166
    1 | 172 | 145 | 95 | 412
    2 | 118 | 124 | 62 | 304
    >2 | 243 | 216 | 114 | 573
In-person on-campus class attendance [Count of Participants; unit: Participants] — Population: Because some participants did not report the characteristic sum of Ns across categories is less than the Overall Number of Baseline Participants.
  Participants
    number analyzed (Participants) | 599 | 548 | 308 | 1455
    0 days/week | 363 | 316 | 67 | 746
    1 day/week | 62 | 51 | 5 | 118
    2-4 days/week | 106 | 107 | 70 | 283
    5 or more days/week | 29 | 30 | 56 | 115
    Not a student | 39 | 44 | 110 | 193
In-person work, volunteer, or on-campus study time [Count of Participants; unit: Participants] — Population: Because some participants did not report the characteristic sum of Ns across categories is less than the Overall Number of Baseline Participants.
  Participants
    number analyzed (Participants) | 599 | 548 | 308 | 1455
    0 days/week | 217 | 192 | 88 | 497
    1 day/week | 75 | 56 | 12 | 143
    2-4 days/week | 207 | 187 | 89 | 483
    5 or more days/week | 100 | 113 | 119 | 332
Member of a fraternity or sorority [Count of Participants; unit: Participants] — Population: Because some participants did not report the characteristic sum of Ns across categories is less than the Overall Number of Baseline Participants.
  Participants
    number analyzed (Participants) | 599 | 548 | 308 | 1455
    Yes | 59 | 68 | 9 | 136
    No | 540 | 480 | 299 | 1319
Current participation in any in-person team sport [Count of Participants; unit: Participants] — Population: Because some participants did not report the characteristic sum of Ns across categories is less than the Overall Number of Baseline Participants.
  Participants
    number analyzed (Participants) | 599 | 548 | 308 | 1455
    Yes | 40 | 44 | 20 | 104
    No | 559 | 504 | 288 | 1351
In last 2 weeks, sat inside a bar, restaurant, cafe, cafeteria [Count of Participants; unit: Participants] — Population: Because some participants did not report the characteristic sum of Ns across categories is less than the Overall Number of Baseline Participants.
  Participants
    number analyzed (Participants) | 599 | 548 | 308 | 1455
    Yes | 400 | 367 | 245 | 1012
    No | 199 | 181 | 63 | 443
In last 2 weeks, usual alcohol consumption [Count of Participants; unit: Participants] — Population: Because some participants did not report the characteristic sum of Ns across categories is less than the Overall Number of Baseline Participants.
  Participants
    number analyzed (Participants) | 599 | 548 | 308 | 1455
    Everyday | 1 | 2 | 5 | 8
    5-6 times per week | 5 | 4 | 5 | 14
    3-4 times per week | 34 | 29 | 19 | 82
    Twice per week | 84 | 75 | 31 | 190
    Once per week | 91 | 69 | 36 | 196
    Once every other week | 94 | 97 | 67 | 258
    None | 290 | 272 | 145 | 707
In last 2 weeks, usual number of drinks when consuming alcohol [Count of Participants; unit: Participants] — Population: Because some participants did not report the characteristic sum of Ns across categories is less than the Overall Number of Baseline Participants.
  Participants
    number analyzed (Participants) | 599 | 548 | 308 | 1455
    7 drinks or more | 3 | 9 | 3 | 15
    4-6 drinks | 54 | 51 | 31 | 136
    1-3 drinks | 250 | 214 | 125 | 589
    Did not drink alcohol | 292 | 274 | 149 | 715
In last 2 weeks, potential exposure to SARS-CoV-2 [Count of Participants; unit: Participants] — Population: Because some participants did not report the characteristic sum of Ns across categories is less than the Overall Number of Baseline Participants.
  Participants
    number analyzed (Participants) | 600 | 548 | 308 | 1456
    No, not to my knowledge | 596 | 534 | 291 | 1421
    Yes, someone with a recent positive test | 4 | 9 | 10 | 23
    Yes, someone with possible symptoms, but no diagnosis or test | 0 | 4 | 3 | 7
    Yes, third party notification system | 0 | 1 | 4 | 5
In last 2 weeks when leaving home, worn a mask inside when around other people [Count of Participants; unit: Participants] — Population: Because some participants did not report the characteristic sum of Ns across categories is less than the Overall Number of Baseline Participants.
  Participants
    number analyzed (Participants) | 599 | 548 | 308 | 1455
    Never | 20 | 23 | 57 | 100
    Rarely | 25 | 29 | 57 | 111
    Occasionally | 48 | 54 | 59 | 161
    Often | 58 | 53 | 38 | 149
    Most of the time | 162 | 153 | 49 | 364
    All of the time | 286 | 236 | 48 | 570
In last 2 weeks when leaving home, maintained physical distancing from others [Count of Participants; unit: Participants] — Population: Because some participants did not report the characteristic sum of Ns across categories is less than the Overall Number of Baseline Participants.
  Participants
    number analyzed (Participants) | 599 | 548 | 308 | 1455
    Never | 9 | 9 | 28 | 46
    Rarely | 24 | 20 | 42 | 86
    Occasionally | 53 | 55 | 77 | 185
    Often | 110 | 96 | 48 | 254
    Most of the time | 243 | 239 | 73 | 555
    All of the time | 160 | 129 | 40 | 329
In last 2 weeks when leaving home, met with others in a group of 10 or more [Count of Participants; unit: Participants] — Population: Because some participants did not report the characteristic sum of Ns across categories is less than the Overall Number of Baseline Participants.
  Participants
    number analyzed (Participants) | 599 | 548 | 308 | 1455
    Never | 273 | 240 | 71 | 584
    Rarely | 188 | 205 | 108 | 501
    Occasionally | 103 | 74 | 69 | 246
    Often | 23 | 23 | 38 | 84
    Most of the time | 3 | 5 | 9 | 17
    All of the time | 9 | 1 | 13 | 23
In last 2 weeks when leaving home, encountered people not wearing masks [Count of Participants; unit: Participants] — Population: Because some participants did not report the characteristic sum of Ns across categories is less than the Overall Number of Baseline Participants.
  Participants
    number analyzed (Participants) | 599 | 548 | 308 | 1455
    Never | 44 | 32 | 7 | 83
    Rarely | 149 | 123 | 18 | 290
    Occasionally | 207 | 205 | 58 | 470
    Often | 110 | 111 | 76 | 297
    Most of the time | 51 | 41 | 74 | 166
    All of the time | 38 | 36 | 75 | 149

OUTCOME MEASURES:

1. Primary Outcome: Efficacy of Moderna COVID-19 Vaccine Against SARS-CoV-2 Infection
Description: Incidence of SARS-CoV-2 infection diagnosed by study PCR among baseline negative participants, with exposure starting from first study PCR and censored at last PCR/outside vaccination and exposure period for the Immediate arm additionally limited to period after the second vaccine dose (period unrestricted for Standard of Care and Vaccine Declined arms: by definition corresponds to unvaccinated exposure). Exact confidence interval.
Time Frame: Measured through Month 4 study visit
Population: Baseline negative with outside vaccination censored incidence rate follow-up
Measure: Number (95% Confidence Interval); unit: events per 100 person years
Units Other Than Participants: person-years
Arm/Group | Immediate Vaccination | Standard of Care | Vaccine Declined
Number analyzed (Participants) | 489 | 531 | 311
Number analyzed (person-years) | 90 | 76 | 50
events per 100 person years | 12.2 [6.1 to 21.9] | 31.8 [20.3 to 47.2] | 89.6 [65.4 to 119.9]
Statistical Analysis 1: Comparison: Immediate Vaccination vs Standard of Care; Cox model on the calendar time scale, stratified by site and adjusted for sex, residence, team sport participation, mask wearing and SARS-CoV-2 exposure risk score. Outside vaccination censoring; Test type: Superiority; Vaccine efficacy, (1-HR) *100% = 52.6, 95% CI 2-sided [-14.1 to 80.3] — "Immediate Vaccination" compared to "Standard of care" (reference). Wald 95% CI

2. Primary Outcome: Effect of Moderna COVID-19 Vaccine on Mean Peak Nasal Viral Load
Description: As a measure of infection and a proxy of infectiousness, mean observed peak viral load (minimum cycle threshold) in nasal samples from FAS-P participants diagnosed with SARS-CoV-2 infection, stratified by lab and target (nucleocapsid gene N1 or N2). Nasal swabs were to be collected daily, and viral load was measured on available specimens taken between the first and last days of PCR-confirmed SARS-CoV-2 infection. Due to early termination, the study was underpowered to look at the vaccine effect on viral load and limited descriptive analysis was performed. The number participants analyzed per row is less than the overall number analyzed as participants were only analyzed by one of the two labs and in few cases the N2 target values could not be measured.
Time Frame: Measured through Month 4 study visit
Population: FAS-P viral load
Measure: Mean (Full Range); unit: Cycle Thresholds
Arm/Group | Immediate Vaccination | Standard of Care | Vaccine Declined
Number analyzed (Participants) | 22 | 23 | 44
Cycle Thresholds
  Lab:Corteva, Target:N1: number analyzed (Participants) | 20 | 17 | 30
  Lab:Corteva, Target:N1 | 25.8 [17.0 to 37.2] | 20.2 [14.6 to 35.8] | 22.3 [12.8 to 37.2]
  Lab:Corteva, Target:N2: number analyzed (Participants) | 20 | 17 | 30
  Lab:Corteva, Target:N2 | 26.3 [17.3 to 38.2] | 20.7 [15.0 to 37.0] | 22.8 [13.2 to 37.5]
  Lab:UW/Northwell, Target:N1: number analyzed (Participants) | 2 | 6 | 14
  Lab:UW/Northwell, Target:N1 | 34.4 [31.3 to 37.5] | 28.8 [18.0 to 39.1] | 24.4 [16.0 to 38.3]
  Lab:UW/Northwell, Target:N2: number analyzed (Participants) | 1 | 6 | 12
  Lab:UW/Northwell, Target:N2 | 34.1 [34.1 to 34.1] | 30.5 [21.1 to 38.6] | 26.2 [18.8 to 34.9]

3. Primary Outcome: Effect of Moderna COVID-19 Vaccine on Median Peak Nasal Viral Load
Description: As a measure of infection and a proxy of infectiousness, median observed peak viral load (minimum cycle threshold) in nasal samples from FAS-P participants diagnosed with SARS-CoV-2 infection, stratified by lab and target (nucleocapsid gene N1 or N2). Nasal swabs were to be collected daily, and viral load was measured on available specimens taken between the first and last days of PCR-confirmed SARS-CoV-2 infection. Due to early termination, the study was underpowered to look at the vaccine effect on viral load and limited descriptive analysis was performed. The number participants analyzed per row is less than the overall number analyzed as participants were only analyzed by one of the two labs and in few cases the N2 target values could not be measured.
Time Frame: Measured through Month 4 study visit
Population: FAS-P viral load
Measure: Median (Inter-Quartile Range); unit: Cycle Thresholds
Arm/Group | Immediate Vaccination | Standard of Care | Vaccine Declined
Number analyzed (Participants) | 22 | 23 | 44
Cycle Thresholds
  Lab:Corteva, Target:N1: number analyzed (Participants) | 20 | 17 | 30
  Lab:Corteva, Target:N1 | 23.9 [21.3 to 29.1] | 19.6 [16.9 to 21.6] | 21.0 [17.3 to 25.9]
  Lab:Corteva, Target:N2: number analyzed (Participants) | 20 | 17 | 30
  Lab:Corteva, Target:N2 | 24.3 [21.9 to 29.5] | 20.0 [17.6 to 22.1] | 21.3 [18.2 to 26.2]
  Lab:UW/Northwell, Target:N1: number analyzed (Participants) | 2 | 6 | 14
  Lab:UW/Northwell, Target:N1 | 34.4 [32.9 to 35.9] | 29.4 [22.8 to 34.6] | 22.5 [19.0 to 29.2]
  Lab:UW/Northwell, Target:N2: number analyzed (Participants) | 1 | 6 | 12
  Lab:UW/Northwell, Target:N2 | 34.1 [34.1 to 34.1] | 31.2 [24.8 to 36.3] | 25.7 [22.1 to 31.1]

4. Secondary Outcome: Efficacy of Moderna COVID-19 Vaccine Against COVID-19 Disease Confirmed by PCR Test and Symptoms
Description: Incidence of study PCR-confirmed SARS-CoV-2 infection and concurrent symptoms captured by daily or weekly symptom reporting (at least one of the following: hospitalization, fever, chills, cough, shortness of breath, difficulty breathing, tiredness/fatigue, muscle aches, joint aches, body aches, headache, change in sense of taste, change in sense of smell, sore throat, nasal congestion, runny nose, nausea, vomiting, diarrhea, oral ulcers and clinical or radiographical evidence of pneumonia) among baseline negative participants. Exposure starting from first study PCR and censored at last PCR/outside vaccination. Participants without concurrent symptom data were assumed not symptomatic and were additionally censored at SARS-CoV-2 infection. Exposure period for the Immediate arm additionally limited to period after the second vaccine dose (period unrestricted for Standard of Care and Vaccine Declined arms: by definition corresponds to unvaccinated exposure). Exact confidence interval.
Time Frame: Measured through Month 4 study visit
Population: Baseline negative with outside vaccination censored incidence rate follow-up
Measure: Number (95% Confidence Interval); unit: events per 100 person years
Units Other Than Participants: person-years
Arm/Group | Immediate Vaccination | Standard of Care | Vaccine Declined
Number analyzed (Participants) | 489 | 531 | 311
Number analyzed (person-years) | 90 | 76 | 50
events per 100 person years | 4.5 [1.2 to 11.4] | 18.5 [10.1 to 31.1] | 53.8 [35.5 to 78.3]
Statistical Analysis 1: Comparison: Immediate Vaccination vs Standard of Care; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; Vaccine efficacy, (1-HR) *100% = 71.0, 95% CI 2-sided [-9.5 to 92.3] — "Immediate Vaccination" compared to "Standard of care" (reference). Wald 95% CI

5. Secondary Outcome: Efficacy of Moderna COVID-19 Vaccine Against SARS-CoV-2 Infection Regardless of Baseline Negativity
Description: Incidence of SARS-CoV-2 infection diagnosed by study PCR among FAS-P participants, with exposure starting from first study PCR and censored at last PCR/outside vaccination and exposure period for the Immediate arm additionally limited to period after the second vaccine dose (period unrestricted for Standard of Care and Vaccine Declined arms: by definition corresponds to unvaccinated exposure). Exact confidence interval.
Time Frame: Measured through Month 4 study visit
Population: FAS-P with outside vaccination censored incidence rate follow-up
Measure: Number (95% Confidence Interval); unit: events per 100 person years
Units Other Than Participants: person-years
Arm/Group | Immediate Vaccination | Standard of Care | Vaccine Declined
Number analyzed (Participants) | 563 | 622 | 452
Number analyzed (person-years) | 103 | 88 | 74
events per 100 person years | 11.7 [6.0 to 20.4] | 28.3 [18.3 to 41.8] | 76.0 [57.4 to 98.7]
Statistical Analysis 1: Comparison: Immediate Vaccination vs Standard of Care; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; Vaccine efficacy, (1-HR) *100% = 41.2, 95% CI 2-sided [-37.7 to 74.9] — "Immediate Vaccination" compared to "Standard of care" (reference). Wald 95% CI

6. Secondary Outcome: Impact of Moderna COVID-19 Vaccine on Secondary Transmission of SARS-CoV-2 Infection
Description: Evaluated by the number of secondary transmission events in close-contact cohorts from main study participants who were SARS-CoV-2 seronegative at enrollment
Time Frame: Measured through Month 4 study visit
Population: Data have not been collected and outcome cannot be reported.
Arm/Group | Immediate Vaccination | Standard of Care | Vaccine Declined
Number analyzed (Participants) | 0 | 0 | 0

7. Secondary Outcome: Efficacy of Moderna COVID-19 Vaccine to Prevent Serologically Confirmed SARS-CoV-2 Infection
Description: Evaluated by SARS-CoV-2 antibodies to the nucleocapsid protein post Month 1 visit among participants who were SARS-CoV-2 seronegative at enrollment
Time Frame: Measured through Month 4 study visit
Population: Data have not been collected and outcome cannot be reported.
Arm/Group | Immediate Vaccination | Standard of Care | Vaccine Declined
Number analyzed (Participants) | 0 | 0 | 0

8. Secondary Outcome: Efficacy of Moderna COVID-19 Vaccine Against COVID-19 Disease Confirmed by PCR Test and Symptoms
Description: Evaluated by SARS-CoV-2 infection confirmed by PCR among participants who were SARS-CoV-2 seronegative at enrollment; reporting at least 2 of the following systemic symptoms: Fever (≥ 38ºC), chills, myalgia, headache, sore throat; or reporting at least one of the following signs/symptoms: cough, shortness of breath or difficulty breathing, new olfactory or taste disorder, clinical or radiographical evidence of pneumonia, thromboembolic event, myocardial infarction, myocarditis, chilblains, or multi-inflammatory syndrome
Time Frame: Measured through Month 4 study visit
Population: Data have not been collected and outcome cannot be reported.
Arm/Group | Immediate Vaccination | Standard of Care | Vaccine Declined
Number analyzed (Participants) | 0 | 0 | 0

9. Secondary Outcome: Effect of Moderna COVID-19 Vaccine on Magnitude of Viral Load Over Time
Description: Summary measures of the viral load curve, all evaluated among participants diagnosed with SARS-CoV-2 infection who were SARS-CoV-2 seronegative at enrollment
Time Frame: Measured through Month 4 study visit
Population: Data have not been collected and outcome cannot be reported.
Arm/Group | Immediate Vaccination | Standard of Care | Vaccine Declined
Number analyzed (Participants) | 0 | 0 | 0

10. Secondary Outcome: Efficacy of Moderna Vaccine Regardless of Baseline Serostatus (SARS-CoV-2 Infection by PCR)
Description: Evaluated by SARS-CoV-2 infection diagnosed by PCR
Time Frame: Measured through Month 4 study visit
Population: Data have not been collected and outcome cannot be reported.
Arm/Group | Immediate Vaccination | Standard of Care | Vaccine Declined
Number analyzed (Participants) | 0 | 0 | 0

11. Secondary Outcome: Effect of Moderna Vaccine on Viral Load Regardless of Baseline Serostatus (Viral Load)
Description: Evaluated by peak viral load in nasal samples from diagnosed participants
Time Frame: Measured through Month 4 study visit
Population: Data have not been collected and outcome cannot be reported.
Arm/Group | Immediate Vaccination | Standard of Care | Vaccine Declined
Number analyzed (Participants) | 0 | 0 | 0

12. Secondary Outcome: Effect of Moderna Vaccine on Secondary Status Regardless of Baseline Serostatus (Secondary Transmission Events)
Description: Evaluated by number of secondary transmission events in close-contact cohorts
Time Frame: Measured through Month 4 study visit
Population: Data have not been collected and outcome cannot be reported.
Arm/Group | Immediate Vaccination | Standard of Care | Vaccine Declined
Number analyzed (Participants) | 0 | 0 | 0

13. Secondary Outcome: Immunogenicity of Moderna COVID-19 Vaccine
Description: Magnitude and response rate of immune responses to vaccination as measured by binding antibody and neutralization assays
Time Frame: Measured through Month 2
Population: Data have not been collected and outcome cannot be reported.
Arm/Group | Immediate Vaccination | Standard of Care | Vaccine Declined
Number analyzed (Participants) | 0 | 0 | 0

14. Secondary Outcome: Immune Responses as Correlates of Risk of SARS-CoV-2 Acquisition, Viral Load, Secondary Infection, and COVID-19 Disease
Description: as for outcome 13
Time Frame: Measured through Month 2
Population: Data have not been collected and outcome cannot be reported.
Arm/Group | Immediate Vaccination | Standard of Care | Vaccine Declined
Number analyzed (Participants) | 0 | 0 | 0

15. Secondary Outcome: Efficacy of Moderna COVID-19 Vaccine Against Asymptomatic SARS-CoV-2 Infection
Description: SARS-CoV-2 infection by PCR or periodic serology
Time Frame: Measured through Month 4 study visit
Population: Data have not been collected and outcome cannot be reported.
Arm/Group | Immediate Vaccination | Standard of Care | Vaccine Declined
Number analyzed (Participants) | 0 | 0 | 0

16. Secondary Outcome: Efficacy of Moderna COVID-19 Vaccine Against SARS-CoV-2 Infection and COVID-19 Disease
Description: SARS-CoV-2 infection diagnosed by PCR among participants who were SARS-CoV-2 seronegative at enrollment and who received all planned immunizations at designated immunization visits
Time Frame: Measured through Month 4 study visit
Population: Data have not been collected and outcome cannot be reported.
Arm/Group | Immediate Vaccination | Standard of Care | Vaccine Declined
Number analyzed (Participants) | 0 | 0 | 0

17. Secondary Outcome: Effect of Moderna COVID-19 Vaccine on Viral Load
Description: Measure of peak viral load among participants who were SARS-CoV-2 seronegative at enrollment and who received all planned immunizations at designated immunization visits
Time Frame: Measured through Month 4 study visit
Population: Data have not been collected and outcome cannot be reported.
Arm/Group | Immediate Vaccination | Standard of Care | Vaccine Declined
Number analyzed (Participants) | 0 | 0 | 0

18. Secondary Outcome: Effect of Moderna COVID-19 Vaccine on Secondary Transmission
Description: Measure of secondary transmission events among participants who were SARS-CoV-2 seronegative at enrollment and who received all planned immunizations at designated immunization visits
Time Frame: Measured through Month 4 study visit
Population: Data have not been collected and outcome cannot be reported.
Arm/Group | Immediate Vaccination | Standard of Care | Vaccine Declined
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: No adverse event information was collected during the study
Description: No adverse event information was collected during the study. Participants were directed to report their adverse events to Vaccine Adverse Event Reporting System (VAERS).
Arm/Group | Immediate Vaccination | Standard of Care | Vaccine Declined
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Informed Consent Form (2021-05-20): https://cdn.clinicaltrials.gov/large-docs/64/NCT04811664/Prot_ICF_000.pdf
  • Statistical Analysis Plan (2023-05-12): https://cdn.clinicaltrials.gov/large-docs/64/NCT04811664/SAP_001.pdf